CLINICAL TRIAL: NCT03256734
Title: Does a Complex Care Discharge Planning Initiative Reduce Unplanned Hospital Readmissions?
Brief Title: Does a Complex Care Discharge Planning Initiative Reduce Unplanned Hospital Readmissions? (G78717-Readmits)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, John Staples, Clinical Assistant Professor, University of British Columbia
Other Study IDs: H17-01039
Record Dates: First submitted 2017-08-18; First posted 2017-08-22 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Patient Readmission

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Policy intervention — Incentive payment for physicians

SUMMARY:
Unplanned hospital readmissions are associated with increases in morbidity, mortality, cost and patient dissatisfaction,. Policymakers continue to seek effective policy solutions to avoid readmissions in order to improve quality of care and reduce unnecessary expenditures,. One attempt to reduce readmissions was implemented on June 1 2012, when the Specialist Services Committee of British Columbia (a partnership of Doctors of BC and the Ministry of Health) introduced the new "G78717" fee code for physicians. The objective of the fee code was to create a financial incentive for physicians to provide a point-of-care supplemental discharge summary to patients and their primary care providers prior to discharge from hospital. Initially, only urgent hospital admissions were eligible for this incentive payment but on Nov 1 2015 the incentive was extended to include elective admissions as well. The other eligibility criteria remained unchanged.

The effectiveness and cost-effectiveness of the fee code intervention is unknown. This study will address important questions relevant to this policy intervention using rigorous methods and empirical data.

This study will employ two methods for measuring changes in readmission risk. First, we will use interrupted (multivariate) time series to measure whether there was a temporal change in provincial readmission risk associated with the implementation of the new fee code.

We will complement the above analyses with a stronger design, comparing hospitalizations for which the fee code was charged (intervention group) with a cohort of clinically similar hospitalizations for which the fee code was not charged (control group). For this approach, multivariate logistic regression will be the primary statistical method. Using this analytic strategy, 30-day readmission risk between the intervention and control group will be measured over time, adjusted for patient-, provider-, and hospitalization-level covariates.

ELIGIBILITY:
Inclusion Criteria:

The study population will be comprised of all hospital discharges in British Columbia between 1 Jan 2002 and 30 June 2017.

Exclusion Criteria:

We will exclude separations with the following International Statistical Classification of Diseases and Related Health Problems, 10th Revision, Canada (ICD-10-CA) codes as the Most Responsible Diagnosis:

* Codes O00 - O99 [Pregnancy, childbirth and the puerperium]
* Codes P00 - P96 [Certain conditions originating in the perinatal period]

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Our study population will be representative of medical and surgical hospital admissions in BC.
  The Interrupted time series (ITS) cohort will be comprised of hospital separations eligible for submission of fee code G78717. We will include all urgent admissions to BC hospitals with discharge dates between 1 Jan 2002 and 30 June 2017 that had a length of stay (LOS) of >4 days and are associated with a specialist Most Responsible Physician (MRP).
  The regression analysis cohort study will be identical to the ITS cohort but will be restricted to index hospitalization discharge dates between 1 Jun 2012 and 31 Jul 2017 (ie. the post-G78717 period).
  The unit of analysis is the index hospital admission (ie. the initial hospital admission of interest). Individual patients can contribute multiple hospital admissions to the cohort over time (although only hospital admissions occurring >30 days after a prior discharge are eligible as index hospital admissions).
Sampling Method: Non-Probability Sample
Enrollment: 300000 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Unplanned hospital readmission within 30 days | 30 days
  Unplanned hospital readmission within 30 days

SECONDARY OUTCOMES:
Unplanned (urgent) hospital readmission within 1 year of index hospital discharge | 1 year
  Unplanned (urgent) hospital readmission within 1 year of index hospital discharge
Primary care visits within 30 days and 1 year of index hospital discharge | 30 days and 1 year
  Primary care visits within 30 days and 1 year of index hospital discharge
Emergency department visit | 30 days and 1 year
  Emergency department visit within 30 days and 1 year of index hospital discharge
Death | 30 days and 1 year
  Death within 30 days and 1 year of index hospital discharge
Use of transitional or stepdown care | 30 days and 1 year
  Use of transitional or stepdown care (eg. rehabilitation, extended care, intermediate /personal care) after discharge from acute care but prior to return home
Improvements in appropriate population-level post-discharge prescription prevalence of an indicated medication | 60 days
  Using health services records, we will identify a sub-cohort of patients with an index admission for acute coronary syndrome, heart failure, or chronic ischemic heart disease. Within this subcohort, we will determine the proportion of patients who filled at least one prescription for beta-blockers within 60 days of index hospital discharge date.
Improvements in appropriate population-level post-discharge prescription prevalence of a contraindicated medication | 60 days
  Using health services records, we will identify a sub-cohort of older adults (aged >/=65 years at date of index hospital discharge date). Within this subcohort, we will determine the proportion of patients who filled at least one prescription for a "potentially inappropriate medication" within 60 days of index hospital discharge date. Our list of "potentially inappropriate medications" has been adapted from those listed in the American Geriatrics Society 2015 Updated Beers Criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Population Data BC, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
Data stewards are legally prohibited from sharing IPD.

REFERENCES:
- [Derived] Staples JA, Yu Y, Khan M, Naik H, Liu G, Brubacher JR, Karimuddin A, Sutherland JM. Physician Financial Incentives to Reduce Unplanned Hospital Readmissions: A Propensity Score Weighted Cohort Study. Am J Med. 2024 Sep;137(9):847-856.e11. doi: 10.1016/j.amjmed.2024.04.042. Epub 2024 May 14. PMID 38750712
- [Derived] Staples JA, Liu G, Brubacher JR, Karimuddin A, Sutherland JM. Physician Financial Incentives to Reduce Unplanned Hospital Readmissions: an Interrupted Time Series Analysis. J Gen Intern Med. 2021 Nov;36(11):3431-3440. doi: 10.1007/s11606-021-06803-8. Epub 2021 May 4. PMID 33948803